CLINICAL TRIAL: NCT06113731
Title: A Randomized, Blinded, Controlled Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of a COVID-19 mRNA Vaccine (ZSVG-02-O) in a Healthy Population 18 Years of Age and Older
Brief Title: A PhaseⅡ Study to Evaluate the Safety and Immunogenicity of COVID-19 Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CNBG-Virogin Biotech (Shanghai) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZSVG-02-O-2022-P2
Record Dates: First submitted 2023-10-31; First posted 2023-11-02 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — CVnCoV COVID-19 vaccine; COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Test vaccine dose 1, 2 dose (Experimental)
  Interventions: Biological: COVID-19 mRNA Vaccine (ZSVG-02-O)
- Test vaccine dose 2, 2 dose (Experimental)
  Interventions: Biological: COVID-19 mRNA Vaccine (ZSVG-02-O)
- Active Comparator, 2 dose (Active Comparator)
  Interventions: Biological: COVID-19 Vaccine (Vero Cell) ,Inactivated
- Test vaccine dose 1, 1 dose (Experimental)
  Interventions: Biological: COVID-19 mRNA Vaccine (ZSVG-02-O)
- Test vaccine dose 2, 1 dose (Experimental)
  Interventions: Biological: COVID-19 mRNA Vaccine (ZSVG-02-O)
- Active Comparator,1 dose (Active Comparator)
  Interventions: Biological: COVID-19 Vaccine (Vero Cell) ,Inactivated

INTERVENTIONS:
Biological: COVID-19 mRNA Vaccine (ZSVG-02-O) — 30 μg
  Arms: Test vaccine dose 1, 1 dose; Test vaccine dose 1, 2 dose
Biological: COVID-19 mRNA Vaccine (ZSVG-02-O) — 60 μg
  Arms: Test vaccine dose 2, 1 dose; Test vaccine dose 2, 2 dose
Biological: COVID-19 Vaccine (Vero Cell) ,Inactivated — COVILO
  Arms: Active Comparator, 2 dose; Active Comparator,1 dose

SUMMARY:
To evaluate the immunogenicity and safety of a COVID-19 mRNA vaccine (ZSVG-02-O) in a healthy population aged 18 years and older.

DETAILED DESCRIPTION:
This study uses a randomized, blinded and controlled design, with age stratification of 18-59 years and ≥60 years , including the test vaccine at different doses (30 μg and 60 μg) and an active control vaccine.

A total of 980 subjects will be enrolled in this study. 490 subjects aged 18-59 years will be randomly assigned to cohort A1 (test vaccine dose 1), A2 (test vaccine dose 2) and A3 (control vaccine) for the 2-dose regimen (0,28-day) and to cohort A4 (test vaccine dose 1), A5 (test vaccine dose 2) and A6 (active control) for the 1-dose regimen in a ratio of 3:3:1:3:3:1. Another 490 subjects aged 60 years or older will be randomized to cohort B1 (test vaccine dose 1), B2 (test vaccine dose 2) and B3 (active control) for the 2-dose regimen (0,28-day), and cohort B4 (test vaccine dose 1), B5 (test vaccine dose 2) and B6 (control vaccine) for the 1-dose regimen in a ratio of 3:3:1:3:3:1.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged ≥18 years of age;
2. Subjects who are in good physical condition as judged by the investigator based on medical history, physical examination and clinical laboratory tests;
3. Subjects who have not been previously vaccinated with a Covid-19 vaccine or who have received the last dose (total dose ≤ 3 doses) of a Covid-19 vaccine at least 6 months ago;
4. Subjects who have not been previously infected with Covid-19, or whose nucleic acid or antigen test has turned negative for more than 3 months after previous Covid-19 infection;
5. Subjects are able to understand the study procedures, have provide written informed consent, and are able to comply with the requirements of the clinical study protocol.

Exclusion criteria

1. Axillary temperature ≥37.3°C;
2. Positive polymerase chain reaction (PCR) test results within the last 48 hours;
3. Women of childbearing potential with a positive urine pregnancy test result, or who are pregnant or breastfeeding, or who have not used effective contraception within 2 weeks prior to enrolment, or women and men who plan to have children within 12 months after full immunisation;
4. History of epilepsy, convulsions or seizures, psychosis or family history of psychosis;
5. Have a history of severe allergy to any medication or vaccination (e.g. acute allergic reaction, urticaria, skin eczema, dyspnoea, angioneurotic oedema, or abdominal pain) or allergy to known components of a Covid-19 vaccine;
6. Have a history of hospital-diagnosed thrombocytopenia or other coagulation disorders;
7. Have a history of hospital-diagnosed known immunological impairment or hypofunction;
8. Subjects who have received whole blood, plasma or immunoglobulin therapy within 3 months;
9. Known or suspected concomitant serious diseases, including: respiratory diseases, acute infections or active chronic diseases, liver and kidney diseases, severe diabetes, malignant tumours, infectious or allergic skin diseases, and HIV infection (with test report);
10. Have serious cardiovascular diseases, cardiopulmonary failure, hypertension that cannot be controlled by medication (systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg on physical examination);
11. Received live attenuated vaccine within 1 month prior to vaccination or other vaccines within 14 days prior to vaccination;
12. Participation in a clinical trial of another drug within 3 months prior to the first dose of vaccine or planning to participate in a clinical trial of another drug during the study period;
13. Any other conditions that the investigator considers inappropriate for participation in this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 980 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titre (GMT) and 4-fold increasing rate of neutralizing antibodies (NAbs) against SARS-CoV-2 on 28 days after full vaccination | 28 days after full immunisation
  Geometric mean titre (GMT) and 4-fold increasing rate of neutralizing antibodies (NAbs) against SARS-CoV-2 on 28 days after full vaccination

SECONDARY OUTCOMES:
GMT and 4-fold increasing rate of NAbs against SARS-CoV-2 on 14 days after full vaccination | 14 days after full immunisation
  GMT and 4-fold increasing rate of NAbs against SARS-CoV-2 on 14 days after full vaccination
GMT and 4-fold increasing rate of NAbs against SARS-CoV-2 on 7 days after the first immunisation | 7 days after the first immunisation
  GMT and 4-fold increasing rate of NAbs against SARS-CoV-2 on 7 days after the first immunisation
Proportion of NAbs against SARS-CoV-2 titres≥1:16, ≥1:32 and ≥1:64 on 14 and 28 days after full immunisation | 14 days and 28 days after full immunisation
  Proportion of NAbs against SARS-CoV-2 titres≥1:16, ≥1:32 and ≥1:64 on 14 and 28 days after full immunisation
GMT, 4-fold increasing rate and ratio of antibody titres ≥1:16, ≥1:32 and ≥1:64 for NAbs against SARS-CoV-2 on 90 and 180 days after full immunisation | 90 days and 180 days after full immunisation
  GMT, 4-fold increasing rate and ratio of antibody titres ≥1:16, ≥1:32 and ≥1:64 for NAbs against SARS-CoV-2 on 90 and 180 days after full immunisation
Incidence and severity of adverse event (AE) within 30 minutes of each dose of vaccination | From the start of each immunisation until 30 minutes after each immunisation
  Incidence and severity of AE within 30 minutes of each dose of vaccination
Incidence and severity of adverse reactions/events 0-14 days after each dose of vaccination | Day 0~Day 14 after each immunisation
  Incidence and severity of adverse reactions/events 0-14 days after each dose of vaccination
Incidence and severity of adverse reactions/events 15-28 days after each dose of vaccination | Day 15~Day 28 after each immunisation
  Incidence and severity of adverse reactions/events 15-28 days after each dose of vaccination
Incidence of serious adverse event (SAE) from the start of vaccination to 12 months after full vaccination | From the first dose of immunisation to 12 months after full immunisation
  Incidence of SAE from the start of vaccination to 12 months after full vaccination

OTHER OUTCOMES:
Changes in cytokine levels in Th1/Th2 cells induced by S protein | From before the first dose of immunisation to 28 days after full immunisation
  Cytokine [IFN-γ, interleukin(IL)-4, IL-2] levels in Th1/Th2 cells changed from pre-dose to 28 days after the full immunisation
Cross-neutralisation against different SARS-CoV-2 variants | From the first dose of immunisation to 28 days after full immunisation
  The cross-neutralization effect of the mRNA vaccine (Omicron strain) against different SARS-CoV-2 variants (ancestral strain, Omicron strain and main circulating strain)

CONTACTS AND LOCATIONS:
Overall Officials: Yunkai Yang, Study Chair — China National Biotec Group Company Limited
Locations (2):
- China (2):
  - Dengfeng Centre for Disease Control and Prevention and Control, Songyang, Henan
  - Henan Provincial Centre for Disease Control and Prevention, Zhengzhou, Henan